CLINICAL TRIAL: NCT00297609
Title: Prevention of Potential Errors in Resuscitation Medications Orders by Means of a Computerized Physician Order Entry With Clinical Decision Support System in Pediatric Critical Care - a Prospective Cohort Study.
Brief Title: Prevention of Errors in Resuscitation Medications Orders by Means of a Computerized Physician Order Entry
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-03-0000-AV-CTIL
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2006-02

CONDITIONS: Critical Care; Pediatrics
Keywords: Resuscitation medication errors; critical care; pediatrics; clinical decision support systems; computerized physician order entry

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Computerized physician order entry with clinical decision support system CPOE+CDSS)completely eliminated errors in filling in the resuscitation medications order forms and significantly reduced time to completing the forms in a pediatric critical care department (PCCD).

DETAILED DESCRIPTION:
Introduction: Computerized physician order entry with clinical decision support system (CPOE+CDSS) is an important tool in attempting to reduce medication errors. The objective of this study was to evaluate the impact of a CPOE+CDSS on (1) the frequency of errors in ordering resuscitation (CPR) medications and (2) the time for printing out the order form, in a pediatric critical care department (PCCD).

Methods: Setting: An 18-bed PCCD in a tertiary-care children's hospital. Design: Prospective cohort study. Measures: Compilation and comparison of number of errors and time to fill in forms before and after implementation of CPOE+CDSS. Errors were identified by reviewing orders and classified as potential adverse drug events (ADEs), medication prescribing errors (MPEs), and rule violations (RVs). They were compared during the year preceding and following implementation of CPOE CDSS. Simulated forms were also used to further test error occurrence. Time to fill in conventional, simulated and CPOE forms was measured and compared.

Results: There were 3 reported incidents of errors among 13,124 CPR medications orders during the year preceding implementation of CPOE+CDSS. These represent errors that escaped the triple check by three independent staff members (two nurses and one physician). There was an average of 11.6 errors/100 orders in the simulated CPR form and potential ADEs occurred at a rate of 11.3/100 orders and MPEs at a rate of 0.3/100 orders. There were no errors after CPOE+CDSS was implemented (100% error reduction). Time to completion of drug forms dropped from 14 min 42 sec to 2 min 14 sec (p<0.001).

Conclusions: CPOE+CDSS completely eliminated errors in filling in the forms and significantly reduced time to completing the form.

ELIGIBILITY:
Inclusion Criteria:

* all admissions to PICU January 2002 - August 2006

Exclusion Criteria:

-

Ages: 3 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vardi, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- PICU SHEBA Medical Center, Tel Litwinsky, Israel